CLINICAL TRIAL: NCT05436340
Title: THE EFFECT OF THE USE OF HEEL PROTECTORS ON THE PREVENTION OF HEEL PRESSURE SORES AND PLANTAR FLEXION CONTRACTURES IN INTENSIVE CARE UNITS
Brief Title: The Effect Of Heel Protector In Intensive Care Units
Acronym: EHePIcu
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Kübra Arslan, Master's Student, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/33-20
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pressure Ulcer, Heel; Plantar Flexion Contracture of Tarsometatarsal Joint
Keywords: Heel Pressure Ulcer; Plantar Flexion Contracture; Heel Protector
MeSH Terms: conditions — Pressure Ulcer | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EHepIcu (Experimental)
  Interventions: Device: The Effect Of Heel Protector In Intensive Care Units; Device: Control group
- Control Grubs (No Intervention)

INTERVENTIONS:
Device: The Effect Of Heel Protector In Intensive Care Units — In the experimental group, foot joint opening and heel pressure sore formation will be observed by using heel protector pad.
  Arms: EHepIcu
Device: Control group — Heel pads will not be used in the control group. Routine maintenance will be applied
  Arms: EHepIcu

SUMMARY:
Purpose: It was aimed to evaluate the effectiveness of using heel protector products for the prevention of heel pressure sore and plantar flexion contracture in patients hospitalized in intensive care units for a long time.

Design: The study is conducted as a Randomized Controlled Study. Method: Heel protectors will be used in the intervention group among the patients in the intensive care unit who meet the inclusion criteria of the study, and the control group will be positioned with a pillow, which is the standard practice. As calculated in the G-Power program with reference to the source, a total of 42 patients were determined to be included in the intervention group and 42 patients in the control group. These patients will be followed for a total of 14 days. Heel Scalp Evaluation and Goniometric Measurements will be made according to Braden Pressure Wound Risk Assessment Scale, Ramsey Sedation Scale, NPUAP and EPUAP Staging System and recorded in the data collection form created by the researcher.

H1: The heel protector is effective in preventing heel pressure ulcer. H0: The heel protector has no effect on preventing heel pressure ulcer. H2: The heel protector is effective in preventing plantar flexion contracture. H0: The heel protector has no effect on preventing plantar flexion contracture. H3: The heel protector is effective in improving the joint range of patients with plantar flexion contracture.

H0: The heel protector has no effect on improving joint range in patients with plantar flexion contracture.

ELIGIBILITY:
Inclusion Criteria:

* High-risk patients; patients who were intubated or extubated in the ICU for at least 5 days and received sedation
* Patients with Braden Pressure Sore Risk Assessment Scale 16 and below
* Patients with a Ramsey Sedation Scale of 4 and above

Exclusion Criteria:

* BMI over 30
* Patients with vascular disease
* Patients with albumin level below 2.5 mg/dL
* Patients mobile within 5 days
* Patients hospitalized with heel pressure ulcer
* Despite being included in the study, the patient becomes mobile before 15 days
* Patients with a medical condition that contraindicates the use of heel protectors

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Foot Joint Opening | for 14 days
  goniometric measurement by the researcher

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat Ateş, Study Director — Üsküdar Üniversitesi
Locations (1):
- Kübra Arslan, Kocaeli, Turkey (Türkiye)